CLINICAL TRIAL: NCT03724227
Title: Expanded Access for ACE-011
Status: No longer available | Type: Expanded Access
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: ACE-011
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2019-10

CONDITIONS: Myelodysplastic Syndrome
Keywords: Expanded Access; Compassionate Use
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — ACE-011

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ACE-011 — ACE-011 will be administered subcutaneous injection
  Other Names: Sotatercept

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to ACE-011.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Celgene, Summit, New Jersey, United States